CLINICAL TRIAL: NCT06213324
Title: Neural Circuit-Specific Mechanisms of Ketamine's Effect on Anhedonia and Anxiety in Depression Using Ultra-High Field 7-Tesla MRI
Brief Title: Neural Circuit Effects of Ketamine in Depression
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James Murrough, Professor of Psychiatry and Neuroscience, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GCO 22-1619; R01MH134045 (NIH)
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Participants in the ketamine arm will receive a single infusion of ketamine
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Participants in the placebo arm will receive a single placebo infusion of normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — 0.5 mg/kg ketamine dissolved in 100 mL saline, delivered intravenously
  Arms: Ketamine
Drug: Placebo — Normal saline delivered intravenously
  Arms: Placebo

SUMMARY:
This project is designed to examine the role of the subgenual anterior cingulate cortex (sgACC) in anhedonia and anxiety in humans with depression, as well as the acute and sustained effects of ketamine on agACC activation and depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

MDD Group

* Male or female aged 18-65 years;
* Ability for participant to comply with the requirements of the study as determined by the PI;
* Capacity to provide informed consent;
* Meets diagnostic criteria for current MDD according to the Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-5);
* In a current major depressive episode (MDE) of at least moderate severity according to DSM-5;
* Women must be using a medically accepted reliable means of contraception (if using an oral contraceptive medication, they must also be using a barrier contraceptive) or not be of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year).
* Women of childbearing potential must have a negative pregnancy test at screening and prior to the infusion.

HC Group

* Male or female aged 18-65 years;
* Capacity to provide informed consent;
* Women must be using a medically accepted reliable means of contraception (if using an oral contraceptive medication, they must also be using a barrier contraceptive) or not be of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year).
* Ability for participant to comply with the requirements of the study as determined by the PI;

Exclusion Criteria:

MDD Group

* Current or history of schizophrenia or other psychotic disorder/episode, bipolar disorder, neurodevelopmental disorder, or neurocognitive disorder;
* Current major depressive disorder with psychotic features;
* Substance use disorder within the past 2 years*;
* Lifetime history of ketamine use disorder;
* Antidepressant medication within 2 weeks of Baseline (4 weeks for fluoxetine);
* Severe current illness as reflected by a CGI score >5;
* Any unstable medical illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease); endocrinologic, neurologic (including history of severe head injury), immunologic, or hematologic disease;
* Clinically significant abnormalities of laboratories, physical examination, or ECG;
* Positive urine toxicology screen for drugs of abuse at the time of screening, except cannabis;
* Women who plan to become pregnant, are pregnant or are breast-feeding (because the medical risk of using ketamine during pregnancy and breast-feeding is unknown);
* Active suicidal intent or plan; CSSRS score >2;
* Any contraindications to MRI, including claustrophobia, any trauma or surgery which may have left magnetic material in the body, magnetic implants or pacemakers, and inability to lie still for 1 hour or more;
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the participant or the quality of the data.

HC Group

* Current or history of any psychiatric, neurodevelopmental disorder, or neurocognitive disorder;
* Substance use disorder within the past 2 years*;
* Any unstable medical illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease); endocrinologic, neurologic (including history of severe head injury), immunologic, or hematologic disease;
* Clinically significant abnormalities of laboratories or physical examination;
* Positive urine toxicology screen for drugs of abuse at the time of screening, except cannabis;
* Current pregnancy;
* Women who are breast feeding;
* Active suicidal intent or plan; CSSRS score >2;
* Any contraindications to MRI, including claustrophobia, any trauma or surgery which may have left magnetic material in the body, magnetic implants or pacemakers, and inability to lie still for 1 hour or more.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
sgACC response to the Incentive Flanker Task | Baseline
  Subgenual anterior cingulate cortex (sgACC) response to reward measured by the BOLD (Blood Oxygen Level Dependent) signal within the sgACC region of the brain, during an fMRI Incentive Flanker Task in healthy controls and in adults with MDD. BOLD signal is the unit of measure of this outcome.

SECONDARY OUTCOMES:
Treatment-related change in sgACC response to the Incentive Flanker Task | Baseline and Day 1
  Treatment-related change from baseline to 1-day post treatment in subgenual anterior cingulate cortex (sgACC) response to reward measured by the BOLD (Blood Oxygen Level Dependent) signal within the sgACC region of the brain, during an fMRI Incentive Flanker Task. MDD adults only.

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD/PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Laurel Morris, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  Any purpose. Specify Other Mechanism Data from this study will be submitted to the National Institute of Mental Health Data Archive (NDA). The NDA is a data repository run by the National Institute of Mental Health (NIMH) that facilitates data sharing across mental health and other research communities. Periodically during and after study completion, the researchers will upload deidentified data information to the NDA. Other researchers nationwide can then file an application to obtain access to deidentified study data for research purposes.
URL: https://nda.nih.gov/